CLINICAL TRIAL: NCT06526260
Title: Very Brief Exposure: Development of a Novel Exposure Modality for Social Anxiety Disorder in Transition-Age Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Bradley Peterson, Chief, Division of Child & Adolescent Psychiatry, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHLA-24-00088; 1R21MH135353-01 (NIH)
Record Dates: First submitted 2024-07-25; First posted 2024-07-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Social Anxiety Disorder
Keywords: Youth; Very Brief Exposure
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Image Exposure Arm (Experimental): Participants will see various images of facial expressions on a computer screen and provide various rating scores about them.
  Interventions: Behavioral: Very Brief Exposure to Facial Expressions

INTERVENTIONS:
Behavioral: Very Brief Exposure to Facial Expressions — In Very Brief Exposure (VBE): a series of rapid micro- exposures to images depicting feared stimuli (e.g., for SAD, judgmental faces). Each image is followed by a masking stimulus to prevent its conscious recognition. This sequence of image-mask stimuli is repeated many times in an exposure session.

SUMMARY:
The goal of this clinical trial is to identify the circuit activations by very brief exposure (VBE) among youth with social anxiety disorder (SAD) in order to develop a novel intervention for those with SAD. The secondary objectives of this study are to measure the effect of VBE on subjective fear ratings, and participants' awareness and tolerance of the exposure stimuli.

* The primary outcome of this study is the mean activation of frontostriatal and prefrontal brain regions to facial stimuli, as measured by Blood Oxygen Level Dependent (BOLD) response, in 4 regions of interest during the magnetic resonance imaging (MRI).
* Another primary outcome of the study is to identify networks of regions subserving emotion regulation and attention, as measured by BOLD response of corresponding brain regions.

Secondary Outcomes

-The secondary outcome of this study is the fear induced by exposure to facial expression stimuli as measured by a 4-point fear scale during the functional magnetic resonance imaging (fMRI) after each block of 10 facial expression stimuli trials.

Participants will participate in an interview where they will answer questions both inside and outside of the MRI scan. Participants will be asked to rate on a scale the imagines they see while undergoing MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Patient Population

  * Males and females aged 16-22. This age range corresponds with our prior studies of very brief exposure (VBE) in Specific Phobia and will include older adolescents while minimizing potential developmental effects on circuit activation.
  * Youth with a Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis of Social Anxiety Disorder (SAD) on Kiddie Schedule for Affective Disorders and Schizophrenia for School-Aged Children, Computerized version (K-SADS-COMP) for youth ages 16-17, or the computerized version of Structured Clinical Interview for the DSM-5 (NetSCID) for youth ages 18+.
* Healthy Population

  • Male and female youth aged 16-22.
* Parents • Parent/caregiver of all ages, no restrictions who are fluent in either English or Spanish.

Exclusion Criteria:

* Patient Population

  * Primary language other than English or Spanish.
  * Active suicidality on the Colombia-Suicide Severity Scale (plan, intent, or behavior)
  * Ferromagnetic implants (e.g., pacemaker), metal braces, retainers, tattoos or permanent make-up with metallic content, transdermal medicinal patches that cannot be removed.
  * Current psychoactive medication.
  * Lifetime diagnosis of: obsessive-compulsive disorder (OCD), psychotic, bipolar, autism spectrum disorder, intellectual disability on the KSADS-COMP or NetSCID.
  * Any serious neurological or medical conditions (e.g., Lupus, cancer, human immunodeficiency virus positive (HIV+)) as reported by potential participants.
  * Current Post-Traumatic Stress Disorder (PTSD) diagnosis.
  * Current severe substance abuse (except tobacco/nicotine).
  * Pregnancy, as determined by the participant's self-report prior to the magnetic resonance imaging (MRI) scan.
* Healthy Population

  * Primary language other than English or Spanish.
  * Lifetime disorders: any anxiety disorders, OCD, psychotic, bipolar, autism spectrum disorder, intellectual disability; any psychiatric disorder in the past 2 years
  * Current depression disorder.
  * Active psychiatric disorder in the past 2 years.
  * Serious neurological or medical conditions.
  * Current psychoactive medication.
  * Ferromagnetic implants (e.g., pacemaker), metal braces, retainers, tattoos or permanent make-up with metallic content, transdermal medicinal patches that cannot be removed.
  * Active suicidality on the Colombia-Suicide Severity Scale (plan, intent, or behavior).
  * Pregnancy, as determined by the participant's self-report prior to the MRI scan.
* Parents • Primary language other than English or Spanish.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mean Activation of Frontostriatal and Prefrontal Brain Regions to disgusted facial expression in Social Anxiety | Day 2
  A hypothesis-driven, group-level analysis will test brain activity, measured as Blood Oxygen Level Dependent (BOLD) response, in 4 regions of interest while minimizing Type II error.
Mean activation of regions subserving emotion, emotion regulation, and attention processing. Mean deactivation of the Default Mode Network. | Day 2
  To identify networks of regions subserving information processing functions, we will employ a voxel-wise, linear mixed model with random- and fixed-effects in group-level analyses. The use of a mixed model with random effects will account for highly discrepant variances between and within participants. We will use Statistical Parametric Mapping 12 Software's (SPM12) implementation of Random Field Theory (RFT) at a voxel-wise level to control for false positives. We will assess the cluster-level statistical significance of task-related brain activity using nonparametric, permutation-based statistical techniques.

SECONDARY OUTCOMES:
Fear induced by exposure to disgusted facial expression in youth with social anxiety as measured by fear scale | Day 2
  After each block of 10 disgusted facial expressions, participants rate levels of fear on a 4-point, 1-4 visual analogue scale with these anchor point: "1 - Minimal fear", "2 - Moderate Fear", "3- Much Fear" and "4 - extreme fear".
Fear induced by exposure to disgusted facial expression in healthy participants as measured by fear scale | Day 2
  After each block of 10 disgusted facial expressions, participants rate levels of fear on a 4-point, 1-4 visual analogue scale with these anchor point: "1 - Minimal fear", "2 - Moderate Fear", "3- Much Fear" and "4 - extreme fear".

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S Peterson, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No